CLINICAL TRIAL: NCT01621607
Title: Gene x Environment Interactions as Risk Factors for Addiction
Brief Title: Individual Differences in Reward and Impulse Control
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999912478; 12-DA-N478
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2017-10-03

CONDITIONS: Drug Addiction; Vulnerability to Substance Addiction
Keywords: fMRI; Monoamines; Environment; Genes; Reward Learning
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Background:

- The risk for becoming addicted to drugs varies among individual, even those using similar drugs in a similar way. It is not known why some people become addicted and others do not. Studies suggest that some genes may increase the risk of addiction. Negative life experiences may also affect the risk of addiction. Researchers want to test smokers and nonsmokers to study genetic and brain function traits that may lead to drug addiction.

Objectives:

- To understand brain function in people who may be at a higher risk of drug addiction.

Eligibility:

* Healthy volunteers between 18 and 55 years of age.
* Smokers (10 to 30 cigarettes per day for more than 2 years) and nonsmokers will be eligible.

Design:

* Participants will be screened with a physical exam and medical history. They will be tested for drug and alcohol use. A blood sample will be collected.
* The study will involve one visit. Participants will have a magnetic resonance imaging (MRI) scan.
* At the visit, participants will answer questions about their health and drug use habits. They will then be trained on the tasks they will do during the MRI scan. After the training, they will have the scan and perform the tasks. The scan and tasks will look at brain function related to rewards and impulsiveness.
* Other computer tests will be given after the scan. These tests will measure learning, memory, and impulsiveness.

DETAILED DESCRIPTION:
Background: Even under similar drug use patterns, the risk for drug addiction varies from individual to individual. However, the neurobiological mechanisms underlying this variability are poorly understood and characterized. Studies suggest that certain traits observed in substance dependent individuals may actually precede drug use, and could augur future substance dependence. Understanding how the presence of these traits increases vulnerability to substance addiction could aid in the development of early intervention, preventative measures, as well as better treatment strategies.

Objective: The primary goal of this protocol is to improve our understanding of increased susceptibility to developing substance addiction. We focus here on particular gene x environment interactions as increased risk factors for substance dependence. The emphasis is on monoaminergic neurotransmitter-related genes thought to influence adaptability to the environment, and, therefore, on cognitive domains related to dopamine and serotonin: reward and punishment learning, and impulse control. To achieve the above objective, the study will be implemented by using cognitive, genetic and neuroimaging testing in adult addicted individuals along with matched controls.

Subject Population: We focus on adult (18-55 years old) smokers and matched non-smoking controls.

Experimental Design: This study involves cognitive, pharmacological and functional magnetic resonance imaging (fMRI) testing in a between-subject design involving neuroimaging and cognitive testing.

Outcome Measures: The primary outcome measures will be BOLD fMRI activation and behavioral performance on various cognitive tasks that deal with impulse control and reward learning, as a function of gene x environment interactions.

ELIGIBILITY:
* INCLUSION CRITERIA FOR ALL PARTICIPANTS:

Between 18 and 55 years old (inclusive);

Must be able to provide informed consent;

Blood pressure (BP) and heart rate (HR) while sitting at or below the following values after five min rest: Systolic BP (SBP) 140 mm Hg, diastolic BP (DBP) 90 mm Hg, heart rate (HR) 100 bpm;

No history of placement in special-education classes as a consequence of serious learning problems (to be assessed during the History and Physical assessment).

Right-handed (based on Edinburgh Handedness Inventory);

Eligible to enter the MRI scanner, as determined though self report on the MRI screening form (from the screening protocol 06-DA-N415).

INCLUSION CRITERIA FOR SMOKERS:

Smoked for at least 2 years, and has generally smoked 10 cpd in the past year and consistently for the past 30 days.

Be able to refrain from smoking for up to 4hrs during the study.

Carry 2 or more plasticity alleles (assessed through protocol # 10-DA-N457 or other IRP protocols)

INCLUSION CRITERIA FOR NON-SMOKERS:

Not have a history of daily cigarette smoking lasting more than a month and no smoking within the past 2 years.

Carry 2 or more plasticity alleles (assessed through protocol # 10-DA-N457 or other IRP protocols)

EXCLUSION CRITERIA FOR ALL PARTICIPANTS:

Report of a history of significant medical/neurological illness that might interfere with imaging data such as HIV positive status, cerebral vascular accident (CVA), central nervous system (CNS) tumor, traumatic brain injury, multiple sclerosis (MS) or other demyelinating diseases, epilepsy, or movement disorders;

History of psychosis or any current DSM-IV axis I disorder (other than simple phobia);

Current use of psychotropic medication that may alter attentional functioning (e.g., Clonidine, antipsychotics, Venlafaxine, stimulants);

Current use of substances on the study visit that might influence performance on tasks as assessed by self-report, carbon monoxide (CO) monitoring, alcohol breathalyzer and urine testing; (and neuromotor evaluation, when needed). If participant is intoxicated at the time of the study visit; he/she will be rescheduled for a later visit.

Meets criteria for abuse, or DSM-IV dependence, or dependence in partial remission, on any drug except nicotine. Past abuse of marijuana or alcohol is acceptable provided it is at least 1 year in the past.

Pregnancy, which will be assessed by history during screening and by urine testing on scan days;

Claustrophobia by self report, or through response to the mock-scanner environment, severe enough to preclude toleration of the scanning environment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2012-06-08; Study Completion 2017-10-03

PRIMARY OUTCOMES:
The primary outcome measures will be BOLD fMRI activation and behavioral performance on various cognitive tasks that deal with impulse control and reward learning, as a function of gene x environment interactions.

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Stein, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

REFERENCES:
- [Background] Barr CS, Newman TK, Lindell S, Shannon C, Champoux M, Lesch KP, Suomi SJ, Goldman D, Higley JD. Interaction between serotonin transporter gene variation and rearing condition in alcohol preference and consumption in female primates. Arch Gen Psychiatry. 2004 Nov;61(11):1146-52. doi: 10.1001/archpsyc.61.11.1146. PMID 15520362
- [Background] Belin D, Mar AC, Dalley JW, Robbins TW, Everitt BJ. High impulsivity predicts the switch to compulsive cocaine-taking. Science. 2008 Jun 6;320(5881):1352-5. doi: 10.1126/science.1158136. PMID 18535246
- [Background] Belsky J, Pluess M. Beyond diathesis stress: differential susceptibility to environmental influences. Psychol Bull. 2009 Nov;135(6):885-908. doi: 10.1037/a0017376. PMID 19883141